CLINICAL TRIAL: NCT04940065
Title: Special Drug-use Surveillance for Kesimpta for s.c. Injection 20 mg Pen (Relapsing-remitting Multiple Sclerosis and Active Secondary Progressive Multiple Sclerosis)
Brief Title: Special Drug-use Surveillance for Kesimpta for s.c. Injection 20 mg Pen
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157G1401
Record Dates: First submitted 2021-06-22; First posted 2021-06-25 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Relapsing-remitting Multiple Sclerosis; Active Secondary Progressive Multiple Sclerosis
Keywords: Kesimpta; multiple sclerosis; Japan
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kesimpta: Patients treated with Kesimpta
  Interventions: Other: Kesimpta

INTERVENTIONS:
Other: Kesimpta — Prospective observational cohort study. There was no treatment allocation.

SUMMARY:
This study was an uncontrolled, central registration system, open-label, multicenter observational study in patients using Kesimpta for the labeled indication.

DETAILED DESCRIPTION:
This was a primary data collection-based special drug-use surveillance to be conducted in accordance with the GPSP ordinance.

Observational period lasted 24 months from the start of treatment with Kesimpta.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written consent to cooperate in this study before the start of treatment with Kesimpta
2. Patients using Kesimpta for the first time for the following indication Indication: prevention of relapses and and prevention of physical disability progression in the following patients

   * Relapsing-remitting MS
   * Active SPMS

Exclusion Criteria:

1. Patients with a history of treatment with a drug containing the same ingredient as Kesimpta (investigational drug or post-marketing clinical study drug)
2. Patients with a history of hypersensitivity to any of the Kesimpta ingredients

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese patients whose registration form is accepted and registration is confirmed.
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 24 months
  An adverse event (AE) is any untoward medical occurrence experienced by a patient administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not related to the medicinal product(s).
Incidence of serious adverse events (SAEs) | 24 months
  A SAE is defined as an adverse event which:
  * Is fatal or life-threatening
  * Results in persistent or significant disability/incapacity
  * Constitutes a congenital anomaly/birth defect
  * Requires inpatient hospitalization or prolongation of existing hospitalization, unless hospitalization is for:
    * Routine treatment or monitoring of the indication under study, not associated with any deterioration in condition
    * Elective or pre-planned treatment for a pre-existing condition that is unrelated to the indication under study and has not worsened since the start of treatment with Kesimpta
    * Social reasons and respite care in the absence of any deterioration in the patient's general condition
  * Is medically significant, i.e., events that jeopardize the patient or may require medical or surgical intervention to prevent one of the outcomes listed above.
Incidence of adverse reactions | 24 months
  An adverse reaction is defined as an adverse event that is suspected by the investigator to be causally related to Kesimpta or whose causality is not recorded.

SECONDARY OUTCOMES:
Physician's Global Assessment | month 12, month 24 (or at treatment discontinuation)
  The investigator comprehensively assessed the symptom changes in relapsing-remitting Multiple Sclerosis (MS) and active Secondary Progressive Multiple Sclerosis (SPMS), rating the changes as "very much improved", "improved", "unchanged", "worsening" or "not assessable" in comparison with the symptoms at the start of this drug, and record the results in the Case report forms (CRFs).
Confirmed disability worsening on Expanded Disability Status Scale (EDSS) | Baseline, month 3, month 6, month 9, month 12, month 15, month 18, month 21, month 24 (or at discontinuation)
  EDSS is a method of quantifying disability in multiple sclerosis (MS) and monitoring changes in the level of disability over time. The scale ranges from 0 (being normal neurological exam and no disability in any functional system) up to 10 (death due to MS). Confirmed disability worsening on EDSS continuing for ≥ 3 months and ≥ 6 months (3mCDW, 6mCDW)
Confirmed improvement on Expanded Disability Status Scale (EDSS) | Baseline, month 3, month 6, month 9, month 12, month 15, month 18, month 21, month 24 (or at discontinuation)
  EDSS is a method of quantifying disability in multiple sclerosis (MS) and monitoring changes in the level of disability over time. The scale ranges from 0 (being normal neurological exam and no disability in any functional system) up to 10 (death due to MS). Confirmed improvement on EDSS continuing for ≥ 6 months (6mCDI)
Number of gadolinium (Gd)-enhancing lesions on Magnetic Resonance Imaging (MRI) | Baseline, month 6, month 12, month 18, month 24 (or at discontinuation)
  The investigator recorded, in the Case report forms (CRFs), the numbers of gadolinium (Gd)-enhancing lesions on MRI
Annual relapse rate | Up to 24 months
  Relapse: Occurrence of new neurological abnormalities or pre-existing neurological abnormalities in stable state or remission occurring at least 30 days after the occurrence of the previous clinical demyelination event that continues at least for 24 hours without pyrexia and infection.
No Evidence of Disease Activity (NEDA-3) | month 12, month 24
  NEDA-3 assessments: no relapse, no new/enlarged MRI lesion, no disability progression on EDSS

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (82):
- Japan (82):
  - Novartis Investigative Site, Ichinomiya, Aichi-ken
  - Novartis Investigative Site, Nagakute, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Tokoname, Aichi-ken
  - Novartis Investigative Site, Toyohashi, Aichi-ken
  - Novartis Investigative Site, Hachinohe, Aomori
  - Novartis Investigative Site, Hirosaki, Aomori
  - Novartis Investigative Site, Chiba, Chiba
  - Novartis Investigative Site, Ichikawa, Chiba
  - Novartis Investigative Site, Narita, Chiba
  - Novartis Investigative Site, Yachiyo, Chiba
  - Novartis Investigative Site, Tōon, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Iizuka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Omuta, Fukuoka
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Fukuyama, Hiroshima
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Hakodate, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Sunagawa, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Mito, Ibaraki
  - Novartis Investigative Site, Tsuchiura, Ibaraki
  - Novartis Investigative Site, Ichinoseki, Iwate
  - Novartis Investigative Site, Morioka, Iwate
  - Novartis Investigative Site, Kagoshima, Kagoshima-ken
  - Novartis Investigative Site, Kanoya, Kagoshima-ken
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Nankoku, Kochi
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Kesennuma, Miyagi
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Nagano, Nagano
  - Novartis Investigative Site, Sasebo, Nagasaki
  - Novartis Investigative Site, Kashihara, Nara
  - Novartis Investigative Site, Tenri, Nara
  - Novartis Investigative Site, Niigata, Niigata
  - Novartis Investigative Site, Ōita, Oita Prefecture
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Fujiidera, Osaka
  - Novartis Investigative Site, Moriguchi, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Kawagoe, Saitama
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Saitama, Saitama
  - Novartis Investigative Site, Wako, Saitama
  - Novartis Investigative Site, Ohtsu, Shiga
  - Novartis Investigative Site, Ōmihachiman, Shiga
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Oyama, Tochigi
  - Novartis Investigative Site, Shimotsuga Gun, Tochigi
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Edogawa City, Tokyo
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Nakano City, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Toyama, Toyama
  - Novartis Investigative Site, Wakayama, Wakayama
  - Novartis Investigative Site, Kudamatsu, Yamaguchi
  - Novartis Investigative Site, Shūnan, Yamaguchi
  - Novartis Investigative Site, Ube, Yamaguchi
  - Novartis Investigative Site, Aomori
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Kobe
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Osaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18382